CLINICAL TRIAL: NCT02063620
Title: The Effect of Different Anesthetic Agents Management on Electrocardiographic Changes of Patients Who Were Operated Under Regional Intravenous Anesthesia
Brief Title: The Effect of Anesthetic Agents Management on ECG Changes of Patients Who Were Operated Under RIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Ilknur Suidiye, assistant professor, Duzce University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: gokceakman; ilknurseker (Other: Duzce University)
Record Dates: First submitted 2014-01-29; First posted 2014-02-14 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Qt Interval, Variation in
Keywords: IVRA, ketamine, lidocaine, ECG
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketamine HCL (Active Comparator): %0.5 Lidocaine+Ketamine HCL 0.8 mg/kg, total 40ml, single dose administration, 30 minute duration, total 200mg lidocaine
  Interventions: Drug: Ketamine HCL
- lidocaine+ serum physiologic (No Intervention): % 0.5 lidocaine+ serum physiologic, total 40ml, total 200 mg lidocaine, 30 minute duration, single dose administration,

INTERVENTIONS:
Drug: Ketamine HCL — ketamine HCL is using as adjuvant agent with local anesthetic agent in regional intravenous anesthesia procedure routinely
  Other Names: Include brande name: ketalar injectable
  Arms: ketamine HCL

SUMMARY:
IVRA can be performed with many local anesthetics and adjuvant agents. Investigators planned to compare cardiac effects and ECG changes by IVRA with lidocaine and lidocaine plus ketamine.

DETAILED DESCRIPTION:
Methods: Patients between 18-60 years, with score of ASA 1-2 and who were undergoing IVRA for short operations on arm and forearm were included. Systolic, diastolic and mean blood pressures, heart rate, SpO2, ECG, adverse effects during the operation were recorded. Double cuffed tourniquet were placed on the extremity to be operated to hinder nerve injuries. Venous blood in the extremity was purged with Esmarch bandage. Proximal cuff was inflated with a pressure 50-100 mmHg higher than systolic blood pressure and the bandage was displaced. Randomly patients were divided into 2 groups. Group 1: %0.5 Lidocaine+Ketamine 0.8 mg/kg; 40 ml. Group 2: %0.5 Lidocaine 40 ml. Anesthetic agent was injected with a rate of 20 ml/min. 20 minutes after injection the distal cuff was inflated and the proximal cuff deflated with a rate of 50 mmHg in every 3 minutes. 0,5,10,15,30,45,60 minutes after the beginning of deflation and 10 minutes after the deflation was completed ECG were recorded. PR,QT,QTc, RR were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18-60 years
2. ASA 1-2 physical status
3. Undergoing IVRA for short operations on arm and forearm

Exclusion Criteria:

1. Allergy to study drugs,
2. Serious cardiac diseases,
3. Respiratory diseases,
4. Renal failure,
5. Drug addiction,
6. Pregnancy,
7. Liver failure,
8. Hypertension,
9. Genetic diseases of musculoskeletal system,
10. Use of antiepileptic drugs, abnormal thyroid functions and operation period over 1 hour.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
QT and QTc intervals | Change QT and QTc intervals from baseline to 60 minutes
  0,5,10,15,30,45,60 minutes after the beginning of deflation and 10 minutes after the deflation was completed ECG were recorded. PR,QT,QTc, RR were recorded.

SECONDARY OUTCOMES:
mean arteryel pressure | Change of mean arteryel pressure from baseline to 60 minutes
  0,5,10,15,30,45,60 minutes after the beginning of deflation and 10 minutes after the deflation was completed

CONTACTS AND LOCATIONS:
Overall Officials: Gokce Akman Kose, Principal Investigator — Duzce University School of Medicine
Locations (1):
- Duzce Univercity Medical Fauculty, Düzce, Turkey (Türkiye)